CLINICAL TRIAL: NCT03877874
Title: The Impact of Anti- Asthmatic Medications on Salivary pH and Dental Caries Pattern in a Group of Egyptian Children With Bronchial Asthma: A Cohort Study
Brief Title: The Impact of Anti- Asthmatic Medications on Salivary pH and Dental Caries Pattern in a Group of Egyptian Children With Bronchial Asthma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Somaya Alaa, Principal investigator, Cairo University
Other Study IDs: 14422017495367
Record Dates: First submitted 2019-03-12; First posted 2019-03-18 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: pH

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Asthmatic children: * Aironyl syrup(Terbutaline sulfate ................. 1.5mg) 0.075-0.29 mg/ kg body weight 3 times daily
  * Apidone syrup(Dexamethone) (0.02 to 0.3 mg per kilogram (kg) of body weight per day, divided and taken 3 or 4 times a day).
  Interventions: Drug: Aironyl syrup(Terbutaline sulfate) + Epidrone syrup(Dexamethone)
- Non-Asthmatic children: no intervention

INTERVENTIONS:
Drug: Aironyl syrup(Terbutaline sulfate) + Epidrone syrup(Dexamethone) — Aironyl syrup(Terbutaline sulfate ................. 1.5mg) 0.075-0.29 mg/ kg body weight 3 times daily Apidone syrup(Dexamethone) (0.02 to 0.3 mg per kilogram (kg) of body weight per day, divided and taken 3 or 4 times a day)
  Groups: Asthmatic children

SUMMARY:
The impact of Anti- Asthmatic medications on salivary pH and dental caries pattern in a Group of Egyptian Children with Bronchial Asthma.

DETAILED DESCRIPTION:
Due to lack of published studies about the impact of anti-asthmatic medications on salivary pH and dental caries pattern among the Egyptian children diagnosed with Bronchial Asthma, this study will be conducted to cover this point.

ELIGIBILITY:
Inclusion Criteria:

* - Children aged 6-12 years old diagnosed with Bronchial asthma (Mixed dentition stage).
* Control group : a matched group aged 6-12 years old
* Patients taking regular medications for the treatment of Bronchial asthma at least for 1 year back
* Both male and female patients will be included.

Exclusion Criteria:

* No other systemic Diseases.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: All patients presented to the Asthma and Allergy Outpatients Clinic of Abu El-Reesh Japanese hospital for kids will be included in the study according to the following criteria.
  -Control group: All patients attending the pediatric dentistry department of faculty of dentistry of Cairo University will be included in the study according to the following criteria.
Sampling Method: Probability Sample
Enrollment: 58 (Estimated)
Dates: Start 2021-07 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
pH of Saliva | 1year
  Digital pH electrode meter

SECONDARY OUTCOMES:
pattern of Dental caries | 1year
  DMFs/defs index

OTHER OUTCOMES:
Drug composition(pH and total sugar content) | 2 minutes
  Digital PH electrode meter